CLINICAL TRIAL: NCT03170596
Title: Microneedling Versus Topical Tazarotene 0.1% Gel for the Treatment of Atrophic Post Acne Scarring - a Randomized Controlled Study
Brief Title: Comparison Between Microneedling Daycare Procedure and Tazarotene 0.1% Gel Local Application in Acne Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Tarun Narang, Assistant Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NK/3486/MD
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Atrophic Post Acne Scarring
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Microneedling procedure will be done on one half of the face and patients will be instructed to apply tazarotene 0.1% gel on the other half of the face
Who Masked: Outcomes Assessor
Masking Description: An independant senior dermatologist who is blinded regarding the modality used for atrophic acne scarring in each half of the face, will be assessing the outcome scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tazarotene gel arm (Experimental): The treatment protocol in this arm will consist of night time application of Tazarotene 0.1% gel during the entire study period. (3 months)
  Interventions: Drug: tazarotene gel 0.1%
- Microneedling arm (Active Comparator): The treatment protocol in this arm will consist of four sessions of microneedling at monthly intervals. (0, 1, 2, 3 months)
  Interventions: Device: Microneedling

INTERVENTIONS:
Drug: tazarotene gel 0.1% — Patients will be instructed to apply 0.1% tazarotene gel as a thin film over the affected area once daily in the evening.
  Arms: Tazarotene gel arm
Device: Microneedling — Microneedling is a method of percutaneous collagen induction
  Arms: Microneedling arm

SUMMARY:
Post acne scarring is a common complication of acne. Cosmetic appearance of the post acne facial scarring can be improved by various methods. Among the procedural methods microneedling (1) is a novel and a promising option. It is a minimally invasive day care procedure for the management of atrophic acne scars. Topical tazarotene 0.1% gel is an effective medical method in the management of acne vulgaris and macular acne scars (2, 3). Based on its mechanism of action and role in collagen synthesis, topical tazarotene is a logical choice to investigate for the management of atrophic post acne scars. This is a pilot study comparing microneedling and topical tazarotene for the treatment of atrophic post acne scarring in regard to extent and rapidity of improvement, patient satisfaction and any adverse events if any.

Thirty six subjects with grade 2 to grade 4 atrophic post acne scars, classified on the basis of Goodman's Qualitative classification (4) criteria will be recruited. Goodman's qualitative and quantitative acne scarring grading system scoring will be performed for the assessment of severity of acne scarring at baseline. The face of each patient will be randomized for monthly microneedling on one side and topical tazarotene 0.1 % gel once a day local application on opposite side, using computer generated random number table. Follow ups will be done at every month until treatment completion (3 months) and 3 months after the last treatment session. Goodman's qualitative and quantitative acne scarring grading system scoring will be performed at 3rd and 6th month follow up visits. An improvement by two grades will be considered as excellent, one grade will be rated as good and no up gradation will be labelled as poor response. Patients will be also assessed by a blinded observer for clinical improvement and scored on a scale of 0 (no improvement) to 10 (maximum) at 3rd and 6th month follow up visits with the help of serial photographs taken under consistent background, position and lighting. All patients will be instructed to assess themselves using Patients' Global Assessment Score 0 (no response) to 10 (maximum) at 3rd and 6th month follow up visits.

The investigators hope the outcome of the present study may propose a newer medical modality for acne scarring, i.e topical tazarotene 0.1% gel, which can be used at home, obviating the need for physician dependant microneedling procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with grade 2 to grade 4 atrophic acne scars, classified on the basis of Goodman's Qualitative classification.6
* Should not have undergone any surgical and/or laser treatment for acne scars in the past 1 year.

Exclusion Criteria:

* Active acne
* History of keloidal tendency/hypertrophic or keloidal scarring on the face due to acne
* Facial scars due to reasons other than acne like varicella, trauma, burns etc
* Collagen vascular disease, bleeding disorders
* Any active bacterial , fungal or viral infection over face
* Pregnant and lactating females
* Known hypersensitivity to tazarotene
* Age less than 18 years
* Patients on anticoagulant therapy or aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Acne scar severity grade at final visit | 6 months
  Change in acne scar severity grade from baseline and at 6 months

SECONDARY OUTCOMES:
Acne scar severity grade at final visit at 3 months | 3 months
  Change in acne scar severity grade from baseline and at 3 months
Patient satisfaction | 6 months
  Patient satisfaction using Patient's global assessment score done at 6 months
Adverse events | 6 months
  Adverse events noted in both arms during the study period of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Narang, MD, Study Chair — Postgraduate Institute of Medical Education and Research, Chandigarh 160012, India
Locations (1):
- Dermatology OPD, New OPD Building, Level 5C, Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doddaballapur S. Microneedling with dermaroller. J Cutan Aesthet Surg. 2009 Jul;2(2):110-1. doi: 10.4103/0974-2077.58529. PMID 20808602
- [Background] Webster GF, Guenther L, Poulin YP, Solomon BA, Loven K, Lee J. A multicenter, double-blind, randomized comparison study of the efficacy and tolerability of once-daily tazarotene 0.1% gel and adapalene 0.1% gel for the treatment of facial acne vulgaris. Cutis. 2002 Feb;69(2 Suppl):4-11. PMID 12095066
- [Background] Phillips TJ, Gottlieb AB, Leyden JJ, Lowe NJ, Lew-Kaya DA, Sefton J, Walker PS, Gibson JR; Tazarotene Cream Photodamage Clinical Study Group. Efficacy of 0.1% tazarotene cream for the treatment of photodamage: a 12-month multicenter, randomized trial. Arch Dermatol. 2002 Nov;138(11):1486-93. doi: 10.1001/archderm.138.11.1486. PMID 12437455
- [Background] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- [Derived] Afra TP, Razmi T M, Narang T, Dogra S, Kumar A. Topical Tazarotene Gel, 0.1%, as a Novel Treatment Approach for Atrophic Postacne Scars: A Randomized Active-Controlled Clinical Trial. JAMA Facial Plast Surg. 2019 Mar 1;21(2):125-132. doi: 10.1001/jamafacial.2018.1404. PMID 30452511